CLINICAL TRIAL: NCT04283344
Title: Evaluation of Demonstrations to End Childhood Hunger - Kentucky
Brief Title: Evaluation of Demonstrations to End Childhood Hunger - KY
Acronym: EDECHKY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Food and Nutrition Service (U.S. Federal Agency)
Collaborators: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG-3198-C-14-0019 (Kentucky)
Record Dates: First submitted 2019-12-12; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Food Insecurity Among Children
Keywords: Food Security; Hunger; Rural; Supplemental Nutrition Assistance Program (SNAP); Food expenditures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KY Ticket to Healthy Food Benefits (Experimental): Households in the treatment group received an extra monthly SNAP benefit amount through two new intervention-related deductions to the SNAP benefit formula: (1) a fixed deduction, depending on county of residence, for transportation costs for six round trips to the grocery store per month; and (2) an earnings deduction equal to 10 percent of earned income for households with at least one employed household member.
  Interventions: Other: KY Ticket to Healthy Food Benefits
- Control Group (No Intervention): Households in the control group continued to receive their regular monthly SNAP benefit amounts.

INTERVENTIONS:
Other: KY Ticket to Healthy Food Benefits — Households in the treatment group received an extra monthly SNAP benefit amount through two new intervention-related deductions to the SNAP benefit formula
  Arms: KY Ticket to Healthy Food Benefits

SUMMARY:
The 2010 Child Nutrition Reauthorization provided funding to test innovative strategies to end childhood hunger and food insecurity. Demonstration projects were funded in Chickasaw Nation, Kentucky, Navajo Nation, Nevada, and Virginia. This study focuses on Kentucky.

Households in the treatment group received an extra monthly SNAP benefit amount through two new intervention-related deductions to the SNAP benefit formula: (1) a fixed deduction, depending on county of residence, for transportation costs for six round trips to the grocery store per month; and (2) an earnings deduction equal to 10 percent of earned income for households with at least one employed household member. Households in the control group continued to receive their regular monthly SNAP benefit amounts.

DETAILED DESCRIPTION:
Objective: To reduce child food insecurity in rural households by raising Supplemental Nutrition Assistance Program (SNAP) benefits to offset higher transportation costs and further strengthen SNAP work incentives.

Target Population: SNAP households with: (1) positive net income, (2) at least one child under the age of 18 by the end of the demonstration period, and (3) living in 17 geographically isolated and poor counties in eastern Kentucky.

Intervention: Households were randomly assigned to either a treatment or control group. Households in the treatment group received an extra monthly SNAP benefit amount through two new intervention-related deductions to the SNAP benefit formula: (1) a fixed deduction, depending on county of residence, for transportation costs for six round trips to the grocery store per month; and (2) an earnings deduction equal to 10 percent of earned income for households with at least one employed household member. Households in the control group continued to receive their regular monthly SNAP benefit amounts.

ELIGIBILITY:
Inclusion Criteria:

* SNAP households with: (1) positive net income, (2) at least one child under the age of 18 by the end of the demonstration period, and (3) living in 17 geographically isolated and poor counties in eastern Kentucky.

Exclusion Criteria:

-

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4504 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Food Insecurity among Children | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 2 or more out of the 8 child-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.

SECONDARY OUTCOMES:
Very Low Food Insecurity among Children | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 5 or more out of the 8 child-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Food Insecurity among Adults | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 3 or more out of the 10 adult-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Household Food Insecurity | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 3 or more out of the 18 items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Food Expenditures | 30 days
  Total amount of Supplemental Nutrition Assistance Program (SNAP) and out-of-pocket food purchases in dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Burke, PhD, Study Director — USDA Food and Nutrition Service

IPD SHARING:
Plan to Share IPD: Yes
Public-use data files are available by request by contacting Michael Burke (michael.burke@usda.gov) or the Office of Policy Support within the USDA Food and Nutrition Service.
Time Frame: April 2019
URL: https://www.fns.usda.gov/ops/evaluation-demonstration-projects-ech

REFERENCES:
- See also: Final Report — https://www.fns.usda.gov/ops/evaluation-demonstration-projects-ech